CLINICAL TRIAL: NCT01903798
Title: A Phase II, Multicenter, Randomized, Open-label Study to Investigate the Safety and Efficacy of Mycophenolate Mofetil and Rilonacept (Anti-interleukin-1) in Patients With Alcoholic Hepatitis
Brief Title: A Safety and Efficacy Study of Mycophenolate Mofetil and Rilonacept in Patients With Alcoholic Hepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: University of Southern California (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); VA Long Beach Healthcare System (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Timothy Morgan, MD, Chief, Hepatology, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAHC Clinical Trial; 1U01AA021886 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Mycophenolic Acid; Prednisolone; rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prednisolone (Lille <0.45) (Active Comparator): At Day 8, after randomization, this participants will continue prednisolone 40 mg/day (current standard of care) for 21 days.
  Interventions: Drug: Prednisolone
- Prednisolone, rilonacept (Lille <0.45) (Experimental): This group will continue Prednisolone (40mg/day). Additionally, they will receive rilonacept (Arcalyst®) once a week for 21 days. After randomization at Day 8, study participants will be given 320 mg subcutaneously (two injections of 2.0 ml, 160 mg each). On Day 15 and Day 22, study participants will be given 160 mg subcutaneously (one injection of 160 mg).
  Interventions: Drug: Prednisolone; Drug: Rilonacept
- Prednisolone (Lille >0.45) (Active Comparator): Prednisolone (40 mg/day) for the first 7 days, after randomization at Day 8, they will stop all therapy.
  Interventions: Drug: Prednisolone
- Prednisolone, mycophenolate(Lille > 0.45) (Experimental): This group will continue Prednisolone (40mg/day). Additionally, they will receive mycophenolate mofetil (CellCept®) for a total of 21 days. After randomization at Day 8, they will receive CellCept® at a dose of 1000 mg per day for the first four days followed by 2000 mg per day (two 500 mg tablets bid) for the remaining 17 days.
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisolone

INTERVENTIONS:
Drug: Mycophenolate mofetil — Immunosuppressive agent
  Arms: Prednisolone, mycophenolate(Lille > 0.45)
Drug: Prednisolone — Corticosteroid
Drug: Rilonacept
  Arms: Prednisolone, rilonacept (Lille <0.45)

SUMMARY:
This clinical trial will test two new therapies for the treatment of alcoholic hepatitis. Patients who "respond" to the current standard of care therapy for alcoholic hepatitis(corticosteroid/prednisolone therapy) after 1 week of treatment will be randomly assigned to either continue on standard therapy, or, to begin treatment with rilonacept in combination with standard therapy. Patients who are "non-responders" to the current standard of care therapy after 1 week of treatment will be randomly assigned to standard of care or to begin treatment with mycophenolate mofetil in combination with standard therapy. Patients will be treated for a total of 4 weeks in this clinical trial. Patients will be followed for up to five months after completing therapy (6 months total).

DETAILED DESCRIPTION:
This is a prospective, randomized trial of two experimental treatments, prednisolone + mycophenolate mofetil and prednisolone + rilonacept, in comparison with standard of care, in patients with alcoholic hepatitis. Patients will start therapy with prednisolone. At Day 8 response to prednisolone will be determined using the Lille score. Patients with a Lille score ≥ 0.45 will be randomized to standard of care (continue prednisolone, stop all therapy and/or offer palliative care) or to have prednisolone continued and mycophenolate added for the next three weeks. Patients with a Lille score <0.45 will be randomized to continue prednisolone alone (standard of care) or to have rilonacept added to their treatment regimen (experimental group) for the next three weeks. Patients will complete follow-up visits at Week 12 and Week 24.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic alcohol consumption (defined as >60g ethanol/day for women and >80g ethanol/day for men) for at least the past 5 years
* Less than 8 weeks between last intake of alcohol and Screening
* Maddrey's Discriminant Function score (DF)>32
* Willing to undergo liver biopsy for histological assessment of alcoholic hepatitis.
* Willing to provide liver tissue, whole blood, stool and ascitic fluid as part of a correlative study
* Onset of jaundice <3 months prior to Screening
* Age greater or equal to 18 years

Exclusion Criteria (Brief):

* Liver disease significantly caused by etiologies other than alcohol.
* Upper GI bleeding requiring transfusion within 48 hours prior to start of prednisolone (Day 1)
* Infection that has been treated with appropriate antibiotics for less than 72 hours or which has not responded appropriately to 72 hours or more of antibiotic treatment prior to start of prednisolone (Day 1)
* Clinical evidence of select active infections in the past 3 months (fungal, mycobacterial, cytomegalovirus (CMV), herpes, coccidioidomycosis, tuberculosis (TB) and human immunodeficiency virus (HIV))
* Renal insufficiency
* Laboratory exclusions
* Hemoglobin <7g/dL
* Total Bilirubin <7.5mg/dL
* Aspartate aminotransferase (AST) >500 IU/mL; or AST:Alanine aminotransferase (ALT) ratio < 1
* Pregnant or breast-feeding or unwilling to use appropriate birth control
* Other clinically significant diseases (uncontrolled diabetes, severe cardiovascular or pulmonary disease, transplant recipient, recent cancer)
* Use of oral or systemic corticosteroids for more than 7 days during the 14 days prior to Day 1 or likely use of oral or systemic corticosteroids in the first 12 weeks of the clinical trial for underlying diseases
* Use of select contraindicated medications
* Previous randomization in the trial
* Based on the investigators judgment, subject is not capable of complying with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R. Morgan, MD, Principal Investigator — VA Long Beach Healthcare System
Locations (3):
- United States (3):
  - VA Long Beach Healthcare System, Long Beach, California
  - LAC USC Medical Center, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 participants were randomized. 3 in the standard of care (with Prednisolone) and 1 in mycophenolate + prednisolone arm. Out of 3 randomized to the SOC arm, 2 had a Lille score of <.45 and one had a Lille score of >.45. The participant who was randomized to mycophenolate + prednisolone had a Lille score of >.45.
Groups:
- Continue Prednisolone (Lille <0.45): Continue prednisolone 40 mg/day (current standard of care) for 21 days.
  Prednisolone: Corticosteroid
- Rilonacept + Prednisolone (Lille <0.45): Prednisolone (40mg/day) and rilonacept (Arcalyst®) subcutaneously once a week for 21 days (320 mg on study Day 8 and 160 mg on study Day 15 and study Day 22).
  Rilonacept: Interleukin-1 blocker
  Prednisolone: Corticosteroid
- Standard of Care (Lille ≥ 0.45): Standard of care therapy (continue prednisolone, stop all therapy and/or offer palliative care)
- Mycophenolate + Prednisolone (Lille ≥ 0.45): Prednisolone (40 mg/day) and mycophenolate mofetil for 21 days (500 mg BID for first 4 days followed by 1000 mg BID for the next 17 days).
  Mycophenolate mofetil: Immunosuppressive agent
  Prednisolone: Corticosteroid
Period: Overall Study
Arm/Group | Continue Prednisolone (Lille <0.45) | Rilonacept + Prednisolone (Lille <0.45) | Standard of Care (Lille ≥ 0.45) | Mycophenolate + Prednisolone (Lille ≥ 0.45)
Started | 2 | 0 | 1 | 1
Completed | 2 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participant was randomized to the Rilonacept + Prednisolone
Groups:
- Total: Total of all reporting groups
Arm/Group | Continue Prednisolone (Lille <0.45) | Rilonacept + Prednisolone (Lille <0.45) | Standard of Care (Lille ≥ 0.45) | Mycophenolate + Prednisolone (Lille ≥ 0.45) | Total
Number analyzed (Participants) | 2 | 0 | 1 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 0 | 3
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.7) |  | 71.2 (0) | 58 (0) | 52 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0 | 0 | 0
  Male | 2 |  | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 0 | 0 | 1
  Not Hispanic or Latino | 1 |  | 1 | 1 | 3
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0
  Asian | 0 |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 1 | 1
  Black or African American | 0 |  | 0 | 0 | 0
  White | 2 |  | 1 | 0 | 3
  More than one race | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day 29 of the Assigned Treatment
Description: To determine whether treatment with prednisolone + mycophenolate mofetil is better than standard of care treatment among patients with alcoholic hepatitis who fail to respond to 1 week of prednisolone (i.e., Lille score of ≥0.45). Primary outcome is survival at Day 29.
  All study participants received the Standard of care (prednisolone) with or without experimental drug at Day 1 (based on randomization). Response to the treatment was determined at Day 8. Data was collected for both responders and non-responders.
Time Frame: Day 8 to Day 29
Population: There was no participant randomized to rilonocept +prednisolone arm
Measure: Count of Participants; unit: Participants
Arm/Group | Continue Prednisolone (Lille <0.45) | Rilonacept + Prednisolone (Lille <0.45) | Standard of Care (Lille ≥ 0.45) | Mycophenolate + Prednisolone (Lille ≥ 0.45)
Number analyzed (Participants) | 2 | 0 | 1 | 1
Participants | 2 | 0 | 1 | 1

2. Secondary Outcome: Number of Patients Reported Ascites
Time Frame: Week 24
Population: No patient was randomized to Rilonacept +prednisolone arm
Measure: Count of Participants; unit: Participants
Arm/Group | Continue Prednisolone (Lille <0.45) | Rilonacept + Prednisolone (Lille <0.45) | Standard of Care (Lille ≥ 0.45) | Mycophenolate + Prednisolone (Lille ≥ 0.45)
Number analyzed (Participants) | 2 | 0 | 1 | 1
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Continue Prednisolone (Lille <0.45) | Rilonacept + Prednisolone (Lille <0.45) | Standard of Care (Lille ≥ 0.45) | Mycophenolate + Prednisolone (Lille ≥ 0.45)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Prednisolone (Lille <0.45) (N=2) | Rilonacept + Prednisolone (Lille <0.45) (N=0) | Standard of Care (Lille ≥ 0.45) (N=1) | Mycophenolate + Prednisolone (Lille ≥ 0.45) (N=1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Prednisolone (Lille <0.45) (N=2) | Rilonacept + Prednisolone (Lille <0.45) (N=0) | Standard of Care (Lille ≥ 0.45) (N=1) | Mycophenolate + Prednisolone (Lille ≥ 0.45) (N=1)
ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other